CLINICAL TRIAL: NCT04329364
Title: A Randomised Controlled Trial Comparing Conventional Open Haemorrhoidectomy and Laser Haemorrhoidoplasty in the Treatment of Symptomatic Haemorrhoids: COHLAH Trial
Brief Title: RCT Comparing Conventional Haemorrhoidectomy With Laser Haemorrhoidoplasty
Acronym: COHLAH
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Collaborators: Biolitec (Unknown)
Responsible Party: Principal Investigator, Koh Hong Xiang Frederick, Associate Consultant, Principal Investigator, Sengkang General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/2930
Record Dates: First submitted 2020-03-19; First posted 2020-04-01 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Hemorrhoids
Keywords: haemorrhoid; laser; haemorrhoidectomy
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: The investigators would be conducting a single-centre RCT simultaneously comparing the conventional open Milligan-Morgan haemorrhoidectomy (COH) and the laser haemorrhoidoplasty procedure (LAH) for the treatment of symptomatic grade ll-lV haemorrhoids.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation is provided through calling the study administrator at time of Examination under Anaesthesia. Thus, the participant is blinded to the procedure. There will also be no cross-over from one study arm to another.
  An independent research administrator, not part of the randomisation process, will also contact the patient 3 months and 1 year after the procedure as mentioned above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Haemorrhoidoplasty (LAH) (Experimental): treatment that we would like to study
  Interventions: Combination Product: Laser Haemorrhoidoplasty (LAH)
- Conventional Open Haemorrhoidectomy (COH) (Active Comparator): gold standard treatment as comparator
  Interventions: Procedure: Open milligan-morgan conventional haemorrhoidectomy

INTERVENTIONS:
Combination Product: Laser Haemorrhoidoplasty (LAH) — Using a laser diode to cause coagulative necrosis to the haemorrhoidal cushion
  Arms: Laser Haemorrhoidoplasty (LAH)
Procedure: Open milligan-morgan conventional haemorrhoidectomy — conventional excisional haemorrhoidectomy
  Arms: Conventional Open Haemorrhoidectomy (COH)

SUMMARY:
Haemorrhoids or piles are the most common colorectal condition in the local population. Patients often present with bleeding with bowel movement or anal discomfort, both of which causes significant anxiety and stress. For symptomatic sizeable piles, the treatment of choice still remains the conventional open excision (COH). However, this technique carries with it a significant risk of bleeding and pain immediately after the operation, leading to some period of discomfort for the patients. The laser haemorrhoidoplasty procedure (LAH) has been shown in preliminary studies to have less pain, and less complications compared to COH. This study aims to directly compare these two techniques in a local Asian population.

The investigators would be conducting a single-centre RCT simultaneously comparing the conventional open Milligan-Morgan haemorrhoidectomy (COH) and the laser haemorrhoidoplasty procedure (LAH) for the treatment of symptomatic grade ll-lV haemorrhoids. Primary outcomes will be post-operative pain while secondary outcomes include post-operative bleeding, readmission and/or reoperations, haemorrhoid-related quality of life (QoL) results and recurrence of symptoms up to a year post procedure

ELIGIBILITY:
Inclusion Criteria:

1. between 21-90 years old
2. presents with symptomatic haemorrhoids as evident from clinical assessment
3. never had any haemorrhoid-related operations performed on them before
4. fit for general anaesthesia
5. able to give informed consent
6. willing to be randomized
7. willing to fill in post-operative questionnaires and be compliant to follow up

Exclusion Criteria:

1. Are pregnant
2. Are prisoners
3. Intellectually, mentally or emotionally deemed not able to provide an informed consent and/or are unable to fill up the post-procedure questionnaires/VAS score
4. Have had previous haemorrhoid procedural treatment before (except Rubber Band Ligation)
5. Declined endoscopic evaluation
6. Are on anti-coagulation
7. Have history of thrombophilia
8. Are on steroids
9. Have haemorrhoids which are incidentally found on endoscopy/clinical examination but are asymptomatic from it

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 10 days from op
  Daily visual analogue pain scale in the first 10 days after surgery. A score of 10 being the worst pain experienced and 1 being no pain experienced.

SECONDARY OUTCOMES:
Operative duration | during operation
  duration of operation
Post-op bleeding | 10 days from operation
  incidence of bleeding post op
readmission | 3 months
  readmission due to complications
recurrence | 1 year post operation
  recurrence of haemorrhoids or symptoms
Quality of Life measures | 10 days, 1 month, 3 months and 1 year post operation
  2 validated questionnaires will be used ([patient self reported symptoms of haemorrhoids] Nystrom, et al. and [standardised haemorrhoidectomy QOL survey] Chew, et al)

CONTACTS AND LOCATIONS:
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
country's personal data protection Act restrictions clearance

REFERENCES:
- [Derived] Koh FH, Foo FJ, Ho L, Sivarajah SS, Tan WJ, Chew MH. Study Protocol for the Use of Conventional Open Haemorrhoidectomy versus Laser Haemorrhoidoplasty in the Treatment of Symptomatic Haemorrhoids: A Randomized Controlled Trial. Eur Surg Res. 2020;61(6):201-208. doi: 10.1159/000513844. Epub 2021 Feb 25. PMID 33631763

DOCUMENTS (2):
  • Study Protocol (2020-03-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT04329364/Prot_000.pdf
  • Informed Consent Form (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT04329364/ICF_001.pdf